CLINICAL TRIAL: NCT03089645
Title: A Phase 1 First Time in Human Study to Evaluate the Safety, Pharmacokinetics and Immunogenicity of MEDI5083 Alone or in Combination With Durvalumab, Tremelimumab, and/or Docetaxel in Advanced Solid Tumors
Brief Title: MEDI5083 Alone and in Combination With Durvalumab, Tremelimumab, and/or Docetaxel.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D6840C00001
Record Dates: First submitted 2017-01-19; First posted 2017-03-24 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — durvalumab; tremelimumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): MEDI5083 monotherapy followed by Durvalumab monotherapy in subjects with advanced solid tumors
  Interventions: Biological: MEDI5083 monotherapy
- Part 2 (Experimental): Sequential MEDI5083 with concurrent Durvalumab or Tremelimumab, and intermittent Medi5083 with concurrent Durvalumab in subjects with advanced solid tumors.
  Interventions: Biological: MEID5083 with Durvalumab or Tremelimumab
- Part 3 (Experimental): Medi5083 with concurrent Durvalumab and Docetaxel randomized against Durvalumab and Docetaxel in subjects with IO refractory/relapsed 2/3L in NSCLC
  Interventions: Biological: Medi5083 with Durvalumab and Docetaxel

INTERVENTIONS:
Biological: MEDI5083 monotherapy — Dose-escalation MEDI5083 monotherapy followed by monotherapy with Durvalumab
  Arms: Part 1
Biological: MEID5083 with Durvalumab or Tremelimumab — Sequential Medi5083 with concurrent Durvalumab or Tremelimumab, and intermittent Medi5083 with concurrent Durvalumab
  Arms: Part 2
Biological: Medi5083 with Durvalumab and Docetaxel — Medi5083 with concurrent Durvalumab and Docetaxel randomized against Durvalumab and Docetaxel
  Arms: Part 3

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics and Immunogenicity of Medi5083 alone or in combination with Durvalumab,Tremelimumab, and/or Docetaxel in adult subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a global Phase 1, first-time-in-human, multicenter, dose-escalation and dose-expansion study of MEDI5083 alone or in combination with Durvalumab, Tremelimumab, and/or Docetaxel.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening or age of consent according to local law
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
3. Histologically or cytologically confirmed metastatic or recurrent tumor types
4. Subjects who have received prior immunotherapy may be eligible
5. Subjects must have at least one measurable lesion
6. Consent to provide archival tumor tissue and pre/on-treatment biopsies
7. Adequate organ and marrow function
8. Consent to use one highly effective method of contraception

Exclusion Criteria:

1. Receipt of any systemic anticancer therapy within 28 days prior to the first dose of MEDI5083
2. Concurrent enrollment in another clinical study
3. Active/prior autoimmune of inflammatory disorders
4. History of immunodeficiency, solid organ transplant, or tuberculosis
5. Known allergy/hypersensitivity to drug or components
6. Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression
7. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of MEDI5083

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) as a measure of safety | From the time of consent through 120 days after last treatment
  Safety Endpoint
Number of participants with Serious Adverse Events (SAEs) as a measure of safety | From the time of consent through 120 days after last treatment
  Safety Endpoint
Number of participants with Dose Limiting Toxicities (DLTs) as a measure of safety | From the time of first dose through 28 days thereafter
  Safety Endpoint
The Maximum Tolerated Dose (MTD) or Highest Protocol-Defined Dose | From the time of first dose through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Safety Endpoint
Discontinuation of investigational products due to toxicity | From the time of first dose through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Safety Endpoint
Clinically significant alterations in vital signs, laboratory parameters, physical examination, and electrocardiogram (ECG) results. | From the time of first dose through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Safety Endpoint
Antitumor activity endpoints OR, based on RECIST v1.1 | Part 3
  Safety Endpoint

SECONDARY OUTCOMES:
Serum MEDI5083 concentration levels | From the time of first dose through 57 days after first treatment
  Pharmacokinetics (PK)
Reduction in peripheral blood CD19+ B cells | From the time of first dose through 57 days after first treatment
  Pharmacodynamics (PD)
Incidence of anti-drug antibody (ADA) responses to MEDI5083 | From the time of first dose through 2 years after last treatment
  Immunogenicity
Objective Response Rate (ORR) | From the time of consent through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Clinical Activity Endpoint
Progression Free Survival (PFS) at 6 months (PFS-6) | From the time of first dose until 6 months after the last subject is dosed
  Clinical Activity Endpoint
Overall Survival (OS) | From the time of consent through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Clinical Activity Endpoint
Disease Control Rate (DCR) | From the time of consent through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Clinical Activity Endpoint
Duration of Response (DoR) | From the time of consent through end of study (2 years after last subject enrolled or earlier at sponsor discretion)
  Clinical Activity Endpoint
Serum Durvalumab concentration levels collected over time | From the time of first dose through 29 days after first treatment
  Pharmacokinetics (PK)
Incidence of anti-drug antibody (ADA) responses to Durvalumab | From the time of first dose through 2 years after last treatment
  Immunogenicity
Incidence of anti-drug antibody (ADA) responses to tremelilumab | From the time of first dose through 2 years after last treatment
  Immunogenicity
Serum tremelimumab concentration levels collected over time | From the time of first dose through 57 days after first treatment
  Pharmacodynamics (PD)
PD of MEDI5083 alone and in combination with Durvalumab and tremelimumab | From the time of first dose through 57 days after first treatment
  Pharmacodynamics (PD)
Safety and tolerability of MEDI5083 with durvalumamb and docetaxel and in subjects with IO relapsed/refractory 2/3L NSCLC | From the time of first dose through 57 days after first treatment
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — Sponsor GmbH
Locations (7):
- United States (4):
  - Research Site, Hackensack, New Jersey
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
- Australia (3):
  - Research Site, Clayton
  - Research Site, Melbourne
  - Research Site, Randwick